CLINICAL TRIAL: NCT05533047
Title: Serum Prostatic Specific Antigen (PSA) Changes After Bipolar and Monopolar Transurethral Resection of the Benign Prostatic Hyperplasia, a Randomized Controlled Study.
Brief Title: Serum Prostatic Specific Antigen Changes After Bipolar and Monopolar TURP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Andrew Hamam Wahba Gerges, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PSA Changes after TURP
Record Dates: First submitted 2022-09-05; First posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: PSA Changes After TURP
MeSH Terms: interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bipolar TURP (Active Comparator): Patients thats will undergo bipolar TURP
  Interventions: Procedure: TURP
- Monopolar TURP (Active Comparator): Patients thats will undergo monopolar TURP
  Interventions: Procedure: TURP

INTERVENTIONS:
Procedure: TURP — Bipolar and monopolar transurethral resection of the benign prostatic hyperplasia

SUMMARY:
To use PSA levels after bipolar and monopolar transurethral resection of the benign prostatic hyperplasia as an indicator of the quality of resection .

DETAILED DESCRIPTION:
PSA is a protein produced from the prostate epithelium and secreted in semen in huge amounts , small amount find its way to the circulation ,its function is to allow mobility of the sperms by interacting with the Semenogelin . clinical BPH can be defined as prostate adenoma/adenomata, causing a varying degree of BOO, which may eventually cause harm to the patients ,Treatment of this condition varies from conservative, medical and surgical depending on factors related to the patient and the surgeon preference . The early reports of minimally invasive treatment of the prostate dated back to 1937, since then and remarkable development is noticed . TURP is the golden treatment in the BPH . Studies compare between the methods according the blood transfusion , operation time retention after catheter removal , urethral complications , TUR syndrome and hospital-stay which show that bipolar is better. To our knowledge after few studies compare between the techniques according PSA also these studies show weakness in their statistically analysis with no difference between the methods .investigators aim is to study the effect of the operations on PSA levels as an indicator of the quality of resection.

ELIGIBILITY:
Inclusion Criteria:

* Patients agreeing to participate, clinically fit, age from 50 to 80 years with LUTS related to benign prostate enlargement with no neurological disorder

Exclusion Criteria:

* Prostate cancer
* Previous urethral or prostate surgery
* Neurogenic bladder
* Urethral stricture
* Patient unfit for surgery

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 2 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
serum PSA changes after bipolar and monopolar transurethral resection of the benign prostatic hyperplasia | within one month after intervention
  To use PSA levels changes after both techniques (bipolar and monopolar transurethral resection of the benign prostatic hyperplasia)as an indicator of the quality of resection

SECONDARY OUTCOMES:
International Prostate Symptom Score | within one month after intervention
  International Prostate Symptom Score after bipolar and monopolar transurethral resection of the benign prostatic hyperplasia

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Elgamal, professor, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Geavlete B, Georgescu D, Multescu R, Stanescu F, Jecu M, Geavlete P. Bipolar plasma vaporization vs monopolar and bipolar TURP-A prospective, randomized, long-term comparison. Urology. 2011 Oct;78(4):930-5. doi: 10.1016/j.urology.2011.03.072. Epub 2011 Jul 29. PMID 21802121
- [Result] Pahwa M, Pahwa M, Pahwa AR, Girotra M, Chawla A, Sharma A. Changes in S-PSA after transurethral resection of prostate and its correlation to postoperative outcome. Int Urol Nephrol. 2013 Aug;45(4):943-9. doi: 10.1007/s11255-013-0474-3. Epub 2013 May 24. PMID 23703547